CLINICAL TRIAL: NCT00890188
Title: The Feasibility of Combing THALIDOMIDE and UFUR in the Treatment of Advanced Colorectal Cancer After Oxaliplatin-Contained Chemotherapy
Brief Title: Thalidomide and Tegafur/Uracil(UFUR) in the Treatment of Advanced Colorectal Cancer
Acronym: UFUR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Peng-Chan Lin/Doctor, National Cheng-Kung University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-97-035
Record Dates: First submitted 2009-04-22; First posted 2009-04-29 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-05

CONDITIONS: Colon Cancer
Keywords: THALIDOMIDE; UFUR; Colorectal cancer; Oxaliplatin
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — Thalidomide; Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- THALIDOMIDE and UFUR (Experimental)
  Interventions: Drug: THALIDOMIDE and UFUR

INTERVENTIONS:
Drug: THALIDOMIDE and UFUR — T: Thalidomide (50): 150 mg/d ((1# tid) U: UFUR(100) 300 mg/d (1# tid) 28 days for one cycle

SUMMARY:
Colorectal cancer is a major health problem in Western society contributing to a high mortality rate. Treatment options for the majority of patients with metastases are limited to cytotoxic chemotherapies. The first line chemotherapy containing with oxaliplatin is recommend by guideline. The use of antiangiogenic agents, either alone or in combination with other therapies may provide an alternative treatment modality in the management of these patients. Metronomic chemotherapy refers to the close, regular administration of a chemotherapeutic drug, over prolonged periods. The advantages of metronomic chemotherapy include reducing acute toxicities and sometimes surprisingly good activity against drug resistant tumors via antiangiogenic effect.

Thalidomide is an agent, which has shown potential in the treatment of hematological and solid tissue malignancies such as multiple myeloma via antiangiogenic mechanism. Tegafur/uracil (UFUR) is one of the effective chemotherapeutics reported to be an effective antiangiogenic agent in an animal model of metastatic colorectal cancers (CRCs).

In the present study, the investigators will try to use low dose metronomic schedule of thalidomide with tegafur/uracil regimen to see the anti tumor efficacy in recurrent and metastasis colorectal cancer patients after oxaliplatin-contained chemotherapy.

The primary endpoints are overall response rate and clinical benefit and the secondary endpoint were to determine the progression free survival, and duration of objective response, the overall survival (OS) and to assess the safety profile. This is a prospective phase II study. After having checked all eligibility criteria, patients will be treated with Tegafur/Uracil (TU) regimen. About 34 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed colorectal carcinoma
* Patients must have received at least one oxaliplatin-contained chemotherapy before the study and did not want to receive or tolerate irinotecan- contained chemotherapy
* Presence of at least one measurable disease which is defined as lesion that can be measured in at least 1 dimension as 20 mm with conventional CT or 10 mm with spiral CT scan
* Age ≥ 18 year, ECOG performance status 0, 1, 2, 3
* White blood cell (WBC) ≥ 3,000/mm3, absolute neutrophil count (ANC) ≥ 1,500/mm3, platelets ≥ 100,000/mm3 and hemoglobin ≥ 8 mg / dl
* Serum creatinine level 2.0 mg/dL or lower
* Serum bilirubin less than 1.5 times the upper limit of normal range (ULN)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) less than 2.5 times the ULN if no demonstrable liver metastases or less than 5 times the ULN in the presence of liver metastases
* Require to wait 28 days before entry onto the study after being treated with any immunotherapy, or biologic systemic (including any target therapy)
* Written informed consent to participate in the trial

Exclusion Criteria:

* Presence of CNS metastasis
* Other malignancy with the exception of curative treated non-melanoma skin cancer or cervical carcinoma in situ within 5 years prior to the entry of study
* Less than 4 weeks since previous treatment
* Concomitant illness that might be aggregated by chemotherapy. For examples, active, non-controlled infection or other active, non-controlled disease such as congestive heart failure, angina pectoris, respiratory insufficiency, arrhythmia. It depends on investigation's decision.
* Women of child-bearing potential without using a reliable and appropriate contraceptive method during study period
* Pre existent sensory or motor neurotoxicity > grade 2 according to National Cancer Institute (NCI) Common Toxicity Criteria (CTC) (disabling paresthesia and/or significant motor loss)
* Patients who are receiving other concomitant chemotherapy, radiotherapy or any other investigational therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Overall response(CR+PR) and Clinical benefit (CR+PR+SD) | 3 months

SECONDARY OUTCOMES:
To determine the progression free survival, overall survival (OS)and assess the safety profile | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Peng Chan Lin, MD, Principal Investigator — National Cheng-Kung University Hospital, Clinical Trial Center
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan